CLINICAL TRIAL: NCT01532960
Title: A Pilot Study of the Immunogenicity of a 9-Peptide Breast Cancer Vaccine Plus Poly-ICLC in Stage I-IV Breast Cancer
Brief Title: Pilot Study of a Breast Cancer Vaccine Plus Poly-ICLC for Breast Cancer
Acronym: Breast 41
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Futility for immune responses to the vaccine. Also, a component of study drug was in short supply.
Sponsor: Craig L Slingluff, Jr (Other)
Responsible Party: Sponsor-Investigator, Craig L Slingluff, Jr, Director, Human Immune Therapy Center, University of Virginia
Organization: University of Virginia (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15881
Record Dates: First submitted 2012-02-08; First posted 2012-02-15 (Estimated); Last update posted 2020-05-08 (Actual); Status verified 2020-05

CONDITIONS: Breast Cancer
Keywords: breast cancer; peptide vaccine; immunotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — poly ICLC

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 9 Peptides from Her-2/neu, CEA, & CTA, peptide-tet, poly-ICLC (Experimental): 9 class I MHC-restricted synthetic peptides (100 mcg each peptide) derived from breast cancer associated proteins, a class II MHC-restricted tetanus derived peptide (200 mcg), plus polyICLC (1 mg).
  Interventions: Biological: poly-ICLC; Biological: 9 Peptides from Her-2/neu, CEA, & CTA; Biological: Peptide-tet

INTERVENTIONS:
Biological: poly-ICLC — poly-ICLC
Biological: 9 Peptides from Her-2/neu, CEA, & CTA — 9 synthetic peptides derived from Her-2/neu, CEA & CTA derived breast cancer proteins.
Biological: Peptide-tet — A class II MHC-restricted helper peptide derived from tetanus toxoid protein.

SUMMARY:
Despite advances in surgical, radiation and medical therapies of early stage breast cancer, some patients will experience disease recurrence. Because recurrence may not happen for years after definitive treatment, there is a period of time between resection and relapse when micrometastatic disease may be amenable to immune eradication or modulation. While the ultimate goal of any cancer treatment is clinical efficacy, the immediate urgency in breast immunotherapy is to define treatments that have immunologic efficacy. In this study, the investigators will determine whether a vaccine consisting of nine-class I breast specific peptides plus a class II tetanus toxoid helper peptide is immunogenic when administered with poly-ICLC to participants with stage IB to IIIA breast cancer in the adjuvant setting.

DETAILED DESCRIPTION:
The study is a single arm, open label, pilot study of safety and immune efficacy of peptide vaccination with poly-ICLC in patients with stage IB-IIIA resected breast cancer. Participants will be patients who have completed their last dose/treatment of any single treatment or combination of adjuvant surgery, radiation, chemotherapy or trastuzumab therapy between 45 days and 6 months (180 days) prior to enrollment.

Each vaccination will be administered on days 1, 8, 15, 36, 57, and 78. All participants will receive 9 class I MHC-restricted synthetic peptides (restricted by HLA-A1, -A2, -A3, or -A31) and a class II MHC-restricted tetanus helper peptide mixed with 1mg poly-ICLC and administered in sterile water. The vaccine will be administered intramuscular (IM) (1 ml) and intradermally (ID) (1 ml) at vaccination sites in the arm and leg. (Each vaccine given IM and ID at one site; site to alternate between arm site opposite the breast cancer and an anterior thigh site.) Participants will be screened for HLA type and must be HLA-A1, -A2, -A3, or -A31 (80% of the Virginia population in prior studies1).

Annual follow-up for progression and survival for 3 years after study withdrawal/completion.

ELIGIBILITY:
Inclusion:

* Patients who have been diagnosed with clinical or pathologic stage I to stage IV adenocarcinoma of the breast (any subtype) who have undergone, and recovered from primary therapy (any combination of surgery, radiation, and/or chemotherapy and/or HER2-directed therapy), with their last dose/treatment (of any single or combination treatment) being between 28 days and 36 months prior to enrollment. Staging will be based on the Seventh Edition AJCC staging system. (Systemic staging with CT or PET scans is not required by AJCC and is not required or exclusionary for this trial).
* Stage IA patients must be high risk based upon triple negative status or HER2+ status
* Patients may or may not be receiving hormonal therapy at the time of study entry.
* Age ≥ 18 years at the time of enrollment
* ECOG performance status of 0 or 1
* Ability and willingness to give informed consent
* HLA-A1, -A2, -A3, or -A31 positive
* Adequate organ function
* HIV and Hepatitis C negative
* Subjects must have a minimum of two intact lymph node basins (any combination of axillary and inguinal basins that have not undergone complete nodal dissection)

Exclusion Criteria

* Known or suspected allergies to any component of the vaccine
* Active infection requiring antibiotics are excluded.
* The following medications or treatments within the 4 weeks (28 days) prior to consenting. These medication and treatments may not be re-started at any time throughout the study in order to remain eligible.

  * Breast tumor resection surgery (reconstructive surgery permitted)
  * Chemotherapy
  * Radiation therapy
  * Allergy desensitization injections
  * Growth factors (e.g., Procrit®, Aranesp®, Neulasta®)
  * Other agents with putative immunomodulating activity (with the exception of non-steroidal anti-inflammatory agents)
  * Any investigational medication
* Tthe following medications or treatments within the 4 weeks (28 days) prior to consenting:

  * Corticosteroids, administered parenterally, orally, or inhaled (Inhaled steroids, such as: Advair®, Flovent®, Azmacort.®)
  * Topical corticosteroids are acceptable.
* Previous vaccination with any of the synthetic peptides included in this protocol.
* Active tuberculosis and not on active antitubercular agents
* Pregnancy.
* Female subjects must not be breastfeeding
* A medical contraindication or potential problem in complying with the requirements of the protocol, in the opinion of the investigator
* New York Heart Association classification as having Class III or IV heart disease
* Stage IV subjects who have anticipated chemotherapy need within the 108 day treatment period for this trial.
* Subjects that have experienced active autoimmune disorders requiring cytotoxic or immunosuppressive therapy within the 6 weeks (42 days) prior to consenting.

  * The following will not be exclusionary:

    * The presence of laboratory evidence of autoimmune disease (e.g., positive ANA titer) without symptoms
    * Clinical evidence of vitiligo
    * Other forms of depigmenting illness
    * Mild arthritis requiring NSAID medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2012-07; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Safety (Frequency of dose limiting adverse events) | 30 days post-administration of the last vaccine
Immune response rate | through day 108
  Measured as the number of IFN-gamma producing cells in the blood in response to the vaccine.

SECONDARY OUTCOMES:
Safety (adverse event profile) | 30 days post-administration of the last vaccine
Immunogenicity- CD8+ T cell specificity | through day 108
  Characterize vaccine specific peripheral CD8+ T-cell specificity by tetramer staining and flow cytometric analysis
Immunogenicity- CD8+ cytokine production | through day 108
  Estimate the Tc1/Tc2 cytokine production bias of circulating vaccine-specific T cells.
Immunogenicity- immue responses among subjects treated with anti-estrogen therapies | through day 108
  Using the ELIspot assay, describe the frequency of immune responses among patients treated with anti-estrogen therapies

CONTACTS AND LOCATIONS:
Overall Officials: Patrick M Dillon, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia Health System, Charlottesville, Virginia, United States

REFERENCES:
- [Derived] Dillon PM, Petroni GR, Smolkin ME, Brenin DR, Chianese-Bullock KA, Smith KT, Olson WC, Fanous IS, Nail CJ, Brenin CM, Hall EH, Slingluff CL Jr. A pilot study of the immunogenicity of a 9-peptide breast cancer vaccine plus poly-ICLC in early stage breast cancer. J Immunother Cancer. 2017 Nov 21;5(1):92. doi: 10.1186/s40425-017-0295-5. PMID 29157306